CLINICAL TRIAL: NCT07259915
Title: Multimodal Prediction of Response to Chemoradiotherapy for Squamous Cell Carcinoma of the Head and Neck
Acronym: MULTINECK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHB24.04
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Squamous Cell Cancer of Head and Neck (SCCHN)
Keywords: multimodal approach; CT DNA; Resonance Magnetic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimodal approach (Experimental): The patient will undergo multimodal imaging and biological sampling
  Interventions: Other: Multimodal approach

INTERVENTIONS:
Other: Multimodal approach — The patient will undergo MRI, PET/can and biological samples

SUMMARY:
The goal of the study lies in offering a multimodal analysis of the post-therapeutic response based on both quantitative parameters and radiomics (CT, MRI, and PET imaging), and on tumor biology, in particular the hypersensitive detection of tumor DNA.

ELIGIBILITY:
Inclusion Criteria:

* Patient with squamous cell carcinoma of the oropharynx (cT2-cT4) or squamous cell carcinoma of the oral cavity (cT2-cT4)
* With lymph node involvement (cN1, cN2, or cN3) (confirmation of lymph node involvement after review of imaging in CCP and without histological confirmation required)
* Eligible for curative treatment with cisplatin-based chemoradiotherapy alone (100 mg/m2 every 3 weeks or 40 mg/m2 weekly)
* Regardless of p16 status
* Affiliated with or covered by a social security system

Exclusion Criteria:

* Head and neck squamous cell carcinomas in other locations (salivary gland, larynx, hypopharynx, cavum, sinuses)
* Primary squamous cell carcinoma of the lymph nodes
* History of radiotherapy to the head and neck region
* Radiochemotherapy not based on the use of cisplatin
* Pregnant or breastfeeding women
* History of invasive cancer in the last 3 years (except for Breslow melanoma less than 1 mm)
* Contraindication to MRI, CT, or PET/CT
* Allergy or contraindication to iodine, gadolinium, or 18F-FDG
* Uncontrolled diabetes (fasting blood glucose greater than 12 mmol/l)
* Patients unable to understand the study for any reason or to comply with the trial requirements (language, psychological, geographical issues, etc.)
* Patients under guardianship or conservatorship
* Patients deprived of their liberty by judicial or administrative decision
* Patients undergoing psychiatric care that renders them incapable of giving their consent
* Patients admitted to a health or social care facility for purposes other than research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Performance of multimodal approach to predict response to chemoradiation | 12 months after treatment
  Estimation of the area under the curve associated with the overall performance of the combined score established by the multimodal approach (PET/CT, MRI, CT, circulating tumor DNA, lymph node tumor DNA) in the post-CRT assessment of the status of a locoregional response within 12 months after chemoradiation.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Universitaire, Rouen

IPD SHARING:
Plan to Share IPD: No